CLINICAL TRIAL: NCT01026233
Title: An Intensive QT/QTc Study to Investigate the Effects of SGN-35 (Brentuximab Vedotin) on Cardiac Ventricular Repolarization in Patients With CD30-Positive Malignancies
Brief Title: Cardiac Safety Study of Brentuximab Vedotin (SGN-35)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-007
Expanded Access: NCT01196208 (No longer available)
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Disease, Hodgkin; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin
Keywords: Antibodies, Monoclonal; Antibody-Drug Conjugate; Antigens, CD30; Disease, Hodgkin; Drug Therapy; Hematologic Diseases; Immunotherapy; Lymphoma; monomethylauristatin E; Lymphoma, Large-Cell, Anaplastic
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin; Hematologic Diseases; Lymphoma | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): brentuximab vedotin
  Interventions: Drug: brentuximab vedotin

INTERVENTIONS:
Drug: brentuximab vedotin — 1.8 mg/kg IV every 21 days
  Other Names: SGN-35

SUMMARY:
The purpose of this study is to evaluate cardiac safety of brentuximab vedotin (SGN-35) in patients with CD30-positive cancers. The study will assess electrical activity of the heart before and after brentuximab vedotin administration. Patients who have stable or improving disease may receive up to 1 year of brentuximab vedotin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory CD30-positive malignancy
* Adequate organ function
* ECOG performance status <2

Exclusion Criteria:

* Cardiac abnormalities (abnormal rhythm, history of significant cardiac event)
* Current diagnosis of primary cutaneous ALCL
* Acute or chronic graft-versus-host disease
* Prior hematopoietic stem cell transplant within specified timeframe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
QTc interval | 2-4 days postdose

SECONDARY OUTCOMES:
ECG parameters | 2-4 days postdose
Blood MMAE levels | Through 4 days postdose
Incidence of proarrhythmic adverse events | Through 1 month following last dose
Incidence of adverse events and laboratory abnormalities | Through 1 month following last dose

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Hunder, MD, Study Director — Seagen Inc.
Locations (9):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Stanford Cancer Center, Stanford, California
  - University of Miami Hospital and Clinics, Miller School of Medicine, Miami, Florida
  - Cardinal Bernardin Cancer Center / Loyola University Medical Center, Maywood, Illinois
  - New York University Cancer Institute, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
- University Hospital of Cologne, Cologne, Germany

REFERENCES:
- [Result] Han TH, Chen R, Advani R, Berryman RB, Smith SE, Forero-Torres A, Rosenblatt JD, Smith MR, Zain J, Hunder NN, Engert A. Brentuximab vedotin does not cause clinically relevant QTc interval prolongation in patients with CD30-positive hematologic malignancies. Cancer Chemother Pharmacol. 2013 Jul;72(1):241-9. doi: 10.1007/s00280-013-2192-z. Epub 2013 May 30. PMID 23719719
- [Derived] Rothe A, Sasse S, Goergen H, Eichenauer DA, Lohri A, Jager U, Bangard C, Boll B, von Bergwelt Baildon M, Theurich S, Borchmann P, Engert A. Brentuximab vedotin for relapsed or refractory CD30+ hematologic malignancies: the German Hodgkin Study Group experience. Blood. 2012 Aug 16;120(7):1470-2. doi: 10.1182/blood-2012-05-430918. Epub 2012 Jul 11. PMID 22786877
- [Derived] Gopal AK, Ramchandren R, O'Connor OA, Berryman RB, Advani RH, Chen R, Smith SE, Cooper M, Rothe A, Matous JV, Grove LE, Zain J. Safety and efficacy of brentuximab vedotin for Hodgkin lymphoma recurring after allogeneic stem cell transplantation. Blood. 2012 Jul 19;120(3):560-8. doi: 10.1182/blood-2011-12-397893. Epub 2012 Apr 17. PMID 22510871